CLINICAL TRIAL: NCT06583174
Title: Evaluation of the Relationship Between Breastfeeding Attitudes and Nutrition Knowledge Levels of Mothers With 0-6 Months Infants
Brief Title: Evaluation of the Relationship Between Breastfeeding Attitudes and Nutrition Knowledge Levels
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2024/07-59
Record Dates: First submitted 2024-08-31; First posted 2024-09-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding
Keywords: Breast milk; breastfeeding; nutrition
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breastfeeding mothers: breastfeeding mothers
  Interventions: Behavioral: Breastfeeding Attitudes

INTERVENTIONS:
Behavioral: Breastfeeding Attitudes — Relationship between Breastfeeding Attitudes and Nutrition Knowledge Levels

SUMMARY:
The importance of breast milk, whose physiological nutritional properties for an infant are not equal to any other food, has been the subject of many studies. In this study, it is aimed to evaluate the relationship between breastfeeding attitude and nutritional knowledge levels of mothers who have 0-6 months infants.

ELIGIBILITY:
Inclusion Criteria:

* volunteering
* Having a baby 0-6 months

Exclusion Criteria:

* not breastfeeding
* Being a pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — breastfeeding mothers
Study Population: breastfeeding mothers
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Nutrition Knowledge | Baseline
  Nutrition Knowledge Scale (NBS): The scale is a 5-point Likert scale with 31 questions. Scale items are scored between 0 and 4 (strongly agree 4 points, strongly disagree 0 points). The highest score that can be obtained from the scale, which is evaluated over the total score, is 126. The higher the score obtained from the scale, the higher the level of nutritional knowledge, and the lower the score, the lower the level of nutritional knowledge.
Breastfeeding Attitude | Baseline
  Breastfeeding Attitude Evaluation Scale: The scale is a 5-point Likert-type scale consisting of 46 items. The total score of the scale is 184. The score of positive items is 88 and the score of negative items is 96. The higher the score, the more positive the breastfeeding attitude is evaluated.
Descriptive assessment | Baseline
  In the general information form of the young individuals participating in the study, demographic information (gender, age, height, body weight, body mass index, etc.) was included.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gökçe İnbaşı, MSc., Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with third parties. The informed consent form has been prepared and approved in this way.